CLINICAL TRIAL: NCT06859450
Title: Local Antibiotic Delivery for Community Acquired Pneumonia - Pilot Study (LANDCAP1)
Brief Title: Local Antibiotic Delivery for Community Acquired Pneumonia
Acronym: LANDCAP-1
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Copenhagen Respiratory Research (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EU-CT: 2024-511413-37-00; 2024-511413-37-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Community Acquired Pneumonia (CAP)
Keywords: Community Acquired Pneumonia; Inhaled levofloxacin; Inhaled antibiotics; feasibility; Chronic obstructive pulmonary disease; asthma; pulmonary healthy; pilot study
MeSH Terms: conditions — Community-Acquired Pneumonia; Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Asthma - Active (Active Comparator): Admitted asthma patient recieving active inhalations
  Interventions: Drug: Levofloxacin
- Asthma - Placebo (Placebo Comparator): Admitted asthma patient recieving placebo inhalations
  Interventions: Drug: Placebo
- Chronic obstructive pulmonary disease - Active (Active Comparator): Admitted COPD-patient recieving active inhalations
  Interventions: Drug: Levofloxacin
- Chronic obstructive pulmonary disease - Placebo (Placebo Comparator): Admitted COPD-patient recieving placebo inhalations
  Interventions: Drug: Placebo
- Pulmonal healthy - Active (Active Comparator): Admitted pulmonary healthy patient recieving active inhalations
  Interventions: Drug: Levofloxacin
- Pulmonal healhty - Placebo (Placebo Comparator): Admitted pulmonary healthy patient recieving placebo inhalations
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levofloxacin — Add-on treatment of inhaled Levofloxacin 240mg twice daily or placebo (saline) twice daily for up to 3 days while admitted.
  Arms: Asthma - Active; Chronic obstructive pulmonary disease - Active; Pulmonal healthy - Active
Drug: Placebo — Add-on treatment of inhaled Levofloxacin 240mg twice daily or placebo (saline) twice daily for up to 3 days while admitted.
  Arms: Asthma - Placebo; Chronic obstructive pulmonary disease - Placebo; Pulmonal healhty - Placebo

SUMMARY:
A randomized, double-blinded clinical pilot study to assess whether addition of inhaled levofloxacin 240 mg twice daily for three days leads to improved or worsened physiological status in CAP patients with and without pre-existing lung disease.

DETAILED DESCRIPTION:
RATIONALE Community-acquired pneumonia (CAP) is a common and potentially severe disease placing a substantial burden on patients and healthcare systems. At the core of the current treatment of CAP is oral or intravenous antibiotics. This poses challenges, both to the individual patient in the form of side-effects due to the antibiotic affecting unintended tissues, as well as to society as current antibiotic prescription patterns may be problematic in the long term due to increasing antimicrobial resistance. Thus, there is a need for alternative treatments that minimize side-effects while reducing the drive of antimicrobial resistance.

The investigators propose inhaled antibiotics as a new treatment modality for CAP. Inhaled administration greatly increases the antibiotic concentration in the lungs, potentially increasing efficacy, while decreasing concentrations in other tissues, potentially reducing side-effects. Especially the gut is important in this regard, as the gut microbiome is much larger than the lung microbiome, therefore the investigators expect that inhaled treatment causes much smaller antibiotic exposure to the bystander bacteria in the gut compared to systemic treatment, reducing antimicrobial resistance selection.

Though results from this study will likely be applicable to other antibiotics, the investigators have specifically chosen to investigate inhaled levofloxacin as it is marketed and has the most favourable side-effect and microbial coverage profile for CAP. Inhaled levofloxacin has been marketed for chronic lung infections since 2015. If the investigators find that inhaled treatment is viable, the investigators hope it will open the path for new inhaled formulations specifically designed for CAP.

To ensure patient safety, the investigators have planned this trial as a small safety trial in which the investigators explore inhaled levofloxacin as an add-on therapy to systemic treatment to collect data on infection control and physiological effects of the drug in a population of CAP patients with or without respiratory comorbidity. These findings will be used in the conduct of a follow-up efficacy trial comparing inhaled treatment to systemic treatment.

The investigators hypothesize that add-on of three days (6 doses over 72 hours) of inhaled levofloxacin to guideline-based treatment of patients with CAP with and without pulmonary comorbidity compared to guideline-based therapy alone is safe and does not cause a worsening of respiratory function defined as decrease in forced end-expiratory volume first second (FEV1).

Further, the investigators hypothesize that such an intervention will lead to comparable disease control defined as an equal number of patients with increasing C-reactive protein, procalcitonin or persistent fever after three days or new onset critical illness.

OBJECTIVES The objective of this study is to determine if addition of inhaled levofloxacin 240 mg twice daily for three days leads to improved or worsened physiological or infectious status in CAP patients with and without pre-existing lung disease.

TRIAL DESIGN A double-blinded randomised controlled trial testing the tolerability and safety of inhaled Levofloxacin in patients admitted to hospital with moderate to severe community-acquired pneumonia.

This study will enrol in total 36 patients:

Of these, all shall have a community-acquired pneumonia (see inclusion criteria below for specific criteria)

Further:

12 subjects with specialist-verified asthma and no other concomitant pulmonary comorbidities.

12 subjects with specialist-verified chronic obstructive pulmonary disease and no other concomitant pulmonary comorbidities.

12 subjects that do not have any pulmonary comorbidities.

INTERVENTION All patients will recieve guideline-based treatment for community-acquired pneumonia. Patients will be randomized 1:1 to recieve blinded add-on treatment with either placebo (saline) or active inhaled levofloxacin 240mg (antibiotic) twice daily for up to 3 days.

All subjects will have the airflow tested before and after their first inhaled treatment and again before discharge or at day 4, whichever comes first.

WORKFLOW Following informed consent, trial participants will fill out a questionnaire about general health status, medicine and comorbidity and the patient's height and weight will be recorded. Furthermore, an electrocardiogram (ECG) will be obtained. For female participants under the age of 55 years who have had a menstruation within 12 months and are not permanently sterile, a pregnancy test will be conducted as part of the screening process. In addition to this, a baseline bedside spirometry will be performed.

The participants will receive a total of 6 inhalations over the course of 72 hours. An investigator or other hospital staff will assist with the medicine administration. Approximately one hour following each inhalation an investigator will perform a clinical assessment of the participant.

SAMPLE SIZE The primary objective of this trial is to evaluate the safety and feasibility of administering inhaled levofloxacin for the treatment of CAP. Additionally the trials aim to gather data and insights to inform the design and implementation of the subsequent main trial (Trial II). To achieve this, the investigators have opted for a conservative patient cohort size. It is recommended to include at least 30 patients in pilot studies, to be able to estimate the standard deviation of population parameters. Therefore, the investigators have chosen to enrol 36 patients stratified by comorbidity in order to ensure robust data collection and analysis.

PUBLICATIONS OF TRIAL RESULTS The results of the trial will be published regardless of whether they are positive, negative, or inconclusive. The trial will be registered and published at clinicaltrials.gov as well as published in an international peer-reviewed scientific journal. Irrespective of the outcome of a clinical trial, within one year from the end of a clinical trial the investigators will submit to the EU database (CTIS) a summary of the results of the clinical trial accompanied by a summary written in a manner that is understandable to laypersons.

If publication in a scientific journal is not possible, the results will be published as an online report.

ETHICAL CONSIDERATIONS Community-acquired pneumonia is a serious and deadly disease which is a great burden on both patients and healthcare systems, and mortality from this condition is still very high. Furthermore, current treatments may not be sustainable in the future due to increasing antimicrobial resistance, which may eventually lead to increasing mortality due to a lack of treatment options.

This study is the first in a line of studies that aims to determine if inhaled antibiotics are a safe, tolerated and an effective way of treatment for a very common and serious disease. Inhaled levofloxacin has been marketed since 2015 and severe adverse events is rare. Overall this study is safe to be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Hospital admission within 24 hours.
2. Radiologically new-onset chest infiltrate that is consistent with pneumonia and symptoms or signs also consistent with pneumonia, such as fever, cough, sputum, dyspnoea and/or chest pain
3. CURB-65 score 3-5
4. C-reactive protein >50 OR central body temperature >38.0 °C (1-2 of these fulfilled)
5. Age ≥ 18 years
6. Able to give informed consent.

Exclusion Criteria:

1. Septic shock according to the sepsis III criteria:41 sequential organ failure assessment (SOFA) score ≥2) and suspected infection (according to attending physician) and persisting hypotension requiring vasopressors to maintain MAP≥65 mmHg and serum lactate level>2 mmol/L (18 mg/dL) despite adequate volume resuscitation (30 mL/kg crystalloid within 3 hours).
2. Oxygen requirement ≥5 L/min to maintain acceptable saturation assessed by the treating physician.
3. Respiratory rate >24/min with relevant oxygen therapy
4. Positive COVID or influenza test (PCR or antigen test)
5. Known allergy to levofloxacin or other fluoroquinolones or a serious adverse reaction when previously treated with a fluoroquinolone, including tendinitis or tendon-rupture related to fluoroquinolone treatment
6. Symptoms of neuropathy (peripheral paraesthesia, hypoesthesia, or hyperalgesia)
7. Known allergy to β-lactam antibiotics or to macrolide antibiotics.
8. Medical history of myasthenia gravis
9. Reduced kidney function (eGFR < 20)
10. Expected transfer to ICU or death within 48 hours or a do not resuscitate ordination at time of recruitment.
11. Suspected aspiration pneumonia, pulmonary abscess, or pleural empyema / complicated parapneumonic effusion.
12. Clinically significant cardiac conduction disorders/arrhythmias or prolonged QTc interval (QTc (f) > 480ms).
13. Pregnancy (a negative pregnancy test is required prior to inclusion of all pre-menopausal women)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-03-04 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in FEV1 after first inhalation from baseline | Enrollment to second assessment - 1 hour
  Proportion of patients with a drop in FEV1 of 20% or 300mL one hour following the first inhalation.

SECONDARY OUTCOMES:
Change in FEV1 from baseline to day 4 or discharge | From baseline to day 4 or discharge. Between 24-72 hours.
  Proportion of patients with a drop in FEV1 of 20% or 300mL from baseline to day 4 or discharge, whichever comes first.
C-reactive protein (CRP) on day 4 higher than any day from baseline to day 3. | Baseline to day 4
  CRP on day 4 higher than on any day from 1 to 3 including baseline.
Physiological status at day 4 | Day 4 assessment
  Mean Arterial Pressure ≤ 65 OR respiratory frequency > 25 OR pulse > 100 OR needing supplemental oxygen (1-4 of these fulfilled) on day 4.
Procalcitonin day 4 compared to any day before including baseline | Baseline to day 4
  Procalcitonin on day 4 higher than on any day from 1 to 3 including baseline.
Temperature at day 4 above 38 degrees celcius | Day 4 assessment
  Temperature ≥ 38.0 °C on day 4.
Patient reported change fra baseline to day 4 | Baseline to day 4
  Patient reported outcome measurements: Changes in Visual Analogue Scales for dyspnoea, cough and fatigue from baseline to day 4. In all of the used scales the value 1 is the lowest meaning "no burden" and a value of 10 meaning "Worst imaginable burden"

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Ulrik S. Jensen, Professor, MD, phD, Study Director — Copenhagen Respiratory Research, Department of Clinical medicine Copenhagen University

IPD SHARING:
Plan to Share IPD: Yes
The results of the trial will be published regardless of whether they are positive, negative, or inconclusive. The trial will be registered and published at clinicaltrials.gov as well as published in an international peer-reviewed scientific journal. Irrespective of the outcome of a clinical trial, within one year from the end of a clinical trial we will submit to the EU database (CTIS) a summary of the results of the clinical trial accompanied by a summary written in a manner that is understandable to laypersons.
  If publication in a scientific journal is not possible, the results will be published as an online report.
Supporting Information: Study Protocol, CSR